CLINICAL TRIAL: NCT04819555
Title: Frequency of SOD1 and C9orf72 Gene Mutations in French ALS
Acronym: GENIALS
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI20-GENIALS
Record Dates: First submitted 2021-03-17; First posted 2021-03-29 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Blood sample; Genetic features
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample for examination of genetic features if required
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adult patients with ALS: incident population of ALS patients followed in the FILSLAN centres.
  Interventions: Genetic: Blood

INTERVENTIONS:
Genetic: Blood — a blood sample will be taken during hospitalisation for diagnostic confirmation or during the quarterly multidisciplinary consultations scheduled as part of the standard follow-up set up for these patients in the ALS centres of the FILSLAN network. If the genetic status is not yet known, this sample will be taken (1 tube of 7mL EDTA) and then sent within 24-48 hours at room temperature to one of the 3 participating molecular biology laboratories according to the criteria defined in the manual of samples being taken in the 3 laboratories.

SUMMARY:
The purpose of the study is to determine the frequency of mutations in the C9orf72 and SOD1 genes in the incident population of ALS patients followed in the FILSLAN centres

DETAILED DESCRIPTION:
After obtaining free and informed consent for genetic characteristic tests, a blood sample will be taken during hospitalisation for diagnostic confirmation or during the quarterly multidisciplinary consultations planned for these patients in the classic follow-up set up within the ALS centres of the FILSLAN network if the genetic status is not already known. This sample will be integrated into the standard management of ALS patients, which includes a neurological examination and paraclinical explorations, including a biological assessment.

The patient will then be reviewed during the standard multidisciplinary follow-up consultations. Information to the patient on his or her C9orf72 or SOD1 genetic status will be included in the quarterly multidisciplinary consultations for the classic follow-up of ALS patients.

It should also be noted that the data (ALSFRS-r score, weight, FEV) collected during the 6 and 12 month consultations will be processed for the purposes of this research.

For patients included in the quarterly multidisciplinary consultations planned in the classic follow-up, if the genetic blood sample was taken during the initial hospitalisation for diagnosis, then it will not be repeated in the framework of the research. In this case, the genetic status of C9orf72 or SOD1 will be available at the inclusion visit and the patient will receive specific information about his or her genetic status.

Consent for the research will nevertheless be obtained in order to have the patient's agreement to the processing of their health data for the purposes of the research at inclusion, 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged ≥ 18 years old
* ALS defined, probable or likely based on neurophysiological data according to Airlie House criteria (Brooks, 2000)
* Sporadic ALS or familial ALS defined by the existence of a case of ALS or FTD among first or second degree relatives of the patient included (Byrne et al, 2011).
* Participant affiliated to a social security scheme
* Free, informed and signed consent for the examination of the genetic characteristics of the participant

Exclusion Criteria:

* All conditions mimicking ALS including motor neuropathies with multiple conduction blocks and all cases of ALS that do not meet the criteria of the Airlie House classification.
* Patients who are cognitively incapable of signing the consent to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: incident population of ALS patients followed in the FILSLAN centres.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
genetic characteristics | Baseline
  frequency of mutations in the C9orf72 and SOD1 genes in the ALS patient population having follow-up for care within the FILSLAN centers French network

SECONDARY OUTCOMES:
neurological examination | 12 months
  describe phenotype of ALS patients according to their genetic status with a neurological examination
ALSFRS-r score | 12 months
  describe homogenous groups of ALS regarding ALSFRS-r score : slope of evolution of the ALSFRS-r score
weight | 12 months
  describe homogenous groups of ALS regarding weight in kg
Expiratory volume | 12 months
  describe homogenous groups of ALS regarding expiratory volume (FEV and LVC) in theoretical %.
Therapeutic management | Baseline
  Calculate the average time elapsed between the request for a molecular diagnosis by the ALS centre and the sending of the result. This will demonstrate the fluidity of the procedure and the ability to quickly inform the patient and the requesting clinician of the genetic status which will be essential to rapidly include patients in targeted gene therapy trials.
Integration of the molecular study into the routine work-up | 12 months
  Compare the percentage of patients who have received genetic analysis to the number of new cases diagnosed in the ALS centres.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe CORCIA, Principal Investigator — University Hospital, Tours
Locations (20):
- France (20):
  - CHU Angers, Angers
  - CHU Bordeaux, Bordeaux
  - CHU de Brest, Brest
  - CHU Lyon, Bron
  - CHU Caen, Caen
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CHU Dijon, Dijon
  - CHU Lille, Lille
  - CHU Limoges, Limoges
  - CHU Marseille, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nancy, Nancy
  - CHU Nice, Nice
  - Paris - Groupe hospitalier de la Pitié Salpetrière, Paris
  - CHU de Rennes, Rennes
  - CHU La Réunion, Saint-Pierre
  - CHU St Etienne, Saint-Priest-en-Jarez
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - University hospital, Tours

IPD SHARING:
Plan to Share IPD: Undecided